CLINICAL TRIAL: NCT01430156
Title: A Randomised Placebo-Controlled Trial to Investigate the Effect of Pre-treatment With Haem Arginate (Normosang) on Heme-Oxygenase 1 (HO-1) Upregulation in Recipients of Deceased Donor Kidneys
Brief Title: Induction of HO-1; a Therapeutic Approach to Reduce Ischaemia Reperfusion Injury (IRI) Following Deceased Donor Renal Transplantation
Acronym: HOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HOT-2011; 2011-004311-23 (EudraCT Number)
Record Dates: First submitted 2011-08-30; First posted 2011-09-07 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Graft Failure; Ischemia-reperfusion Injury
Keywords: Renal Transplantation; Ischemia-reperfusion injury; Heme-oxygenase 1; Heme arginate
MeSH Terms: conditions — Reperfusion Injury | interventions — heme arginate; Hemin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Heme arginate (Normosang) (Active Comparator): This arm will receive 2 doses of Heme Arginate (trade name Normosang); 1 dose prior to transplant and another on day 2. This is a product derived from human hemin and has been used for over 20 years in clinical practice with few side-effects.
  Interventions: Drug: Heme arginate (Normosang)
- 0.9% saline (Placebo Comparator): The saline will be given as an IV infusion in the same manner as the Heme Arginate (active comparator) infusion.
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Heme arginate (Normosang) — 3mg/kg as a single IV infusion prior to transplant over 30 mins and same dose repeated on day 2 post-transplantation. Each drug infusion will be followed by 100ml saline IV to flush the line.
  Other Names: Heme Arginate; Hemin
  Arms: Heme arginate (Normosang)
Drug: 0.9% sodium chloride — Solution for infusion, this will be given prior to transplantation and again on day 2; the same as active drug.
  Other Names: Normal saline
  Arms: 0.9% saline

SUMMARY:
This is a blinded, placebo-controlled, randomised controlled trial looking at the effects of Heme arginate (HA) on cadaveric renal transplantation. The investigators know that HA can upregulate HO-1, which has been shown to have a protective effect on animal transplants.

The investigators will be giving HA/placebo to participants prior to transplant and repeat again on day 2 post-transplant and compare outcomes.

DETAILED DESCRIPTION:
Patients will be recruited from the East of Scotland transplant waiting list and consent when they arrive in the hospital. The investigators will randomise them to drug or placebo and give the infusion prior to induction for their transplant.

A blood sample will be taken prior to infusion and a renal biopsy will be taken before the graft is implanted. These will be used as baseline values.

Patients will receive standard care from our unit. The investigators will use the routine blood test results (urea and creatinine) to determine the function of the graft.

The investigators will take blood samples 24 hours after infusion of drug/placebo and use this to determine the primary outcome. Blood tests will be taken daily and a renal biopsy taken on day 5 to fulfil secondary objectives.

ELIGIBILITY:
Inclusion Criteria:

* all patients receiving a cadaveric single kidney transplant
* patients on a standard immunosuppressive regime

Exclusion Criteria:

* patients on different immunosuppressives
* patients receiving 3rd or subsequent kidney transplant
* patients are fully anti-coagulated
* patients unable to take Heme Arginate
* patients unable to give informed consent
* patients on combined anti-platelet agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Macrophage/monocyte HO-1 protein levels | 24 hours
  We will measure the level of HO-1 protein in isolated macrophages/ monocytes in a peripheral blood sample taken at 24 hours after drug infusion

SECONDARY OUTCOMES:
Macrophage/monocyte HO-1 mRNA levels | 24 hours
  We will measure HO-1 mRNA levels in macrophages/monocytes from a peripheral blood sample taken at 24 hours.
HO-1 protein in kidney transplant | 5 days
  We will measure the level of HO-1 protein in kidney tissue from a biopsy sample taken 5 days after drug infusion. This will be compared to baseline
Effect on transplanted kidney function | daily for 5 days
  We will record how the kidney functions by determining presence or absence of delayed graft function.
Urinary biomarkers as markers of injury | daily for 5 days
  We will collect urine to measure the presence of specific urinary biomarkers and correlate with renal function.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna Marson, MD, Study Director — Senior Lecturer, Transplant Surgery, University of Edinburgh; Rachel Thomas, MBChB, Principal Investigator — Clinical Research Fellow, University of Edinburgh; Stephen McNally, PhD, Principal Investigator — University of Edinburgh; David Kluth, PhD, Principal Investigator — University of Edinburgh
Locations (1):
- Royal Infirmary of Edinburgh/ University of Edinburgh, Edinburgh, Lothian, United Kingdom

REFERENCES:
- [Derived] Thomas RA, Czopek A, Bellamy CO, McNally SJ, Kluth DC, Marson LP. Hemin Preconditioning Upregulates Heme Oxygenase-1 in Deceased Donor Renal Transplant Recipients: A Randomized, Controlled, Phase IIB Trial. Transplantation. 2016 Jan;100(1):176-83. doi: 10.1097/TP.0000000000000770. PMID 26680374